CLINICAL TRIAL: NCT04023279
Title: Effects of Myofascial Release of the Brachial Biceps and TENS Over the Elbow Pain, Hand Prehensile Strength and Functionality of Superior Extremity in Women With Symptomatology of Chronic Lateral Epicondylalgia
Brief Title: Effects of Myofascial Release and TENS Over Pain, Hand Prehensile Strength and Functionality of Superior Extremity in Women With Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda Merino Alvarez (Other)
Responsible Party: Sponsor-Investigator, Fernanda Merino Alvarez, Sponsor and Principal Investigator Fernanda Merino Alvarez, Universidad Nacional Andres Bello
Organization: Universidad Nacional Andres Bello (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UniversidadNAB
Record Dates: First submitted 2019-07-07; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Musculoskeletal Manipulations
Keywords: Manual therapy; Myofascial release; Lateral epicondylitis; Transcutaneous electrical nerve stimulation; Pain; Strength; Functionality
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Transcutaneous Electric Nerve Stimulation; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Quantitative, experimental prospective, explanatory type, randomized controlled parallel with simple blind.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The hidden assignment of the participants was carried out using the method of opaque envelopes sealed and numbered consecutively.
  The assessor in charge of evaluating the participants was blind to the treatment assignment, where he proceeded to take the measurements with a prior instruction of the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): Conventional TENS of 100 Hz and 100 usec for 20 minutes
  Interventions: Other: TENS
- Myofascial Therapy (Experimental): Conventional TENS of 100 Hz and 100 usec for 20 minutes plus myofascial release therapy in the brachial biceps; Seven to fifteen transverse sliding repetitions and three repetitions of longitudinal sliding
  Interventions: Other: TENS; Other: Myofascial therapy

INTERVENTIONS:
Other: TENS — 100 Hz and 100 usec for 20 minutes
  Other Names: Transcutaneous electrical nerve stimulation
Other: Myofascial therapy — Seven to fifteen transverse sliding repetitions and three repetitions of longitudinal sliding of myofascial release therapy
  Arms: Myofascial Therapy

SUMMARY:
This study evaluated the additive effect of myofascial release therapy on the brachial biceps on conventional management (TENS) in pain intensity, hand prehensile strength and upper limb functionality of individuals with lateral epicondylalgia.

DETAILED DESCRIPTION:
This study determined the additive effect of the myofascial release therapy of brachial biceps on TENS in the variables pain intensity, hand prehensile strength and upper limb functionality of individuals with lateral epicondylalgia, compared to a group that received only TENS. This was done in a sample of 32 individuals, assigned in two groups: group A that received an application of TENS and group B that received an application of TENS plus myofascial release therapy.

Contrary to the hypothesis, the application of myofascial release therapy added to the application of TENS proved to generate a significant change only in the prehensile hand force with respect to the group that received only TENS.

ELIGIBILITY:
Inclusion Criteria:

* Female between 30 and 50 years old.
* Belong to the administrative staff of the university in question
* Have a symptomatic diagnosis of chronic lateral epicondylitis (> 6 weeks)

Exclusion Criteria:

* Being pregnant
* Have done moderate or intense aerobic or anaerobic sport activities of any kind 72 hours before the registrations
* Have an orthopedic, rheumatologic, neuropsychiatric or associated comorbidities diagnosed.
* Have suffered a fracture or trauma involving the upper extremity 4 months before the intervention.
* Be in medical, pharmacological or kinesthetic treatment during the intervention or 2 weeks before this.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity numerical rating scale | One month
  Self-reported measure of pain intensity. It consists on asking to assess pain intensity by selecting a number on a scale of 11 horizontal points. It is represented from 0 (without pain) to 10 (the worst possible pain) A score of 1 to 4 indicates mild pain; 5-6, moderate pain; and 7 to 10, severe pain.
Pressure pain threshold | Immediately after treatment
  Is the minimum pressure that induces pain or discomfort. It was measured with a algometer. It is expressed in units of pressure as kilograms per square centimeter per second (Kg / cm2 / s).
Prehensile hand strength | Immediately after treatment
  It is the ability to compress the hand, related to the functional integrity of the upper extremity as an index of general health. It was measured with a dynamometer. It was measured according to the criteria established by the American Society of Hand Therapists. It is measured in kilograms
Change in Elbow functionality. | One month
  Functionality is a generic term that includes bodily functions, body structures, activities and participation. It shows the positive aspects of a person's interaction and the context. It was obtained through a scale of functionality (Oxford Elbow Score), which is composed of three domains (subscales); elbow, pain and social-psychological function, which underlie 12 questions, which are internally consistent, one-dimensional and do not have redundancy of items.
  The scores of each domain are calculated as the sum of the score of each individual element, where each case is expressed on a scale from 0 to 100 where, a score of 0.84 indicates a substantial improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Fuentes, PhD, Study Director — Universidad Andres Bello
Locations (1):
- Universidad Andres Bello, Talcahuano, Concepción, Chile